CLINICAL TRIAL: NCT05423405
Title: Efficacy of Acupressure in Depression as Non-invasive Nursing Intervention - a Randomized Single-blind Trial With Psychological and Physiological Criteria
Brief Title: The Efficacy of Acupressure Therapy on Patient With Depression
Acronym: Akupress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Psychiatric Clinics Basel (Network)
Responsible Party: Principal Investigator, Hamdy Shaban, Principal Investigator, University Psychiatric Clinics Basel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Akupressur-Therapie
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Depressive Disorder; Depressive Disorder, Major; Depressive Symptoms
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Patients population with depression (mild, moderate, or severe)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): Treatment as usual with pharmacotherapy and other complementary therapies
- Sham (Sham Comparator): No actual acupoint pressed but same settings as in acupressure therapy
  Interventions: Other: Acupressure
- Intervention (Experimental): Treatment as usual plus acupressure intervention with selected acupoints pressure
  Interventions: Other: Acupressure

INTERVENTIONS:
Other: Acupressure — selected acupoint pressure
  Other Names: TCM
  Arms: Intervention; Sham

SUMMARY:
A new nursing intervention with non-invasive acupressure protocol for activation of parasympathetic nervous system to reduce stress related depression symptoms.

DETAILED DESCRIPTION:
Acupressure is a treatment method in which manual pressure is applied to specific points or areas of the body. According to the principles of Traditional Chinese Medicine (TCM), these acupuncture points are stimulated along the energy channels (meridians) of the body. Finger pressure is mainly used here, in some cases also with a relaxing massage. According to TCM, this can stimulate the energy flow of the Qi. The therapist also tries to treat energetic blockages. Acupuncture is recommended for psychological problems, pain syndromes and sleep disorders, among other things.

Acupressure has been established as an additional therapy offer in private department J of the UPK since the beginning of 2021. Patients with depression and anxiety disorders subjectively benefit from the treatment in terms of reducing stress symptoms and improving relaxation.

Although patient acceptance is high, there are no high-quality studies on accompanying acupressure as part of standard treatments for depression, anxiety or sleep disorders. Their effectiveness in psychiatric patients is therefore controversial. Although there are few studies from "Western medicine" institutions, most of the clinical studies were carried out by Chinese colleagues. In most cases, only subjective assessment instruments were used to assess effectiveness without evaluating objective biomarker measurements such as cortisol concentration, brain-derived neurotrophic factor (BDNF) or cytokines.

A hypothesis on the effectiveness of acupressure in western medicine has not been established. The vagus nerve stimulation may play a role and thus the activation of the parasympathetic nervous system - which in turn could lead to a reduction in stress symptoms and an increase in relaxation and regeneration in the short and/or medium term. The role of the social bonding hormone oxytocin has not been studied so far.

The aim of this study is to evaluate the efficacy of acupressure adjunctive therapy in Major Depressive Disorder (MDD) as part of evidence-based treatment as usual (TAU) as a randomized, single-blind study.

Physiological and psychological assessment instruments should be used: cortisol levels in the saliva; serum oxytocin and BDNF levels; Heart rate variability, Hamilton Depression Rating Scale (HAM-D; third-party rating scale) and Beck Depression Inventory-II (BDI-II, self-rating scale).

The acupressure therapy protocol specially developed in the UPK could thus be established as a non-invasive, non-drug nursing therapy tool and achieve scientifically sound application in the UPK and other clinics, provided that proof of effectiveness is achieved.

We are pursuing a long-term strategy with our study because we are convinced that the current treatment options for depression are not sufficient and could be supplemented and improved by innovative and complementary therapies. Acupuncture can play a helpful role as an easily accessible and inexpensive method.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Primary diagnosis of MDD with a current moderate-to-severe episode (HAM-D score > 16) 55
* Treatment as usual for depression
* Able to read and understand study procedures and participant's information
* Agree to receive acupressure therapy

Exclusion Criteria:

* Suicidal ideation
* Antipsychotic medication
* Primary diagnosis other than MDD
* Contradiction for acupressure (skin diseases, pregnancy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline self reported Depression Severity | with 2 month
  Beck Depression Inventory BDI (Max score >40 High depression, Min score < 10 Normal)
Change from Baseline Depression Severity | with 2 month
  Hamilton Depression Rating Scale HDRS (Max score >18 Severe (moderate) depression, Min < 7 no depression)

SECONDARY OUTCOMES:
Change from baseline heart rate | with 2 month
  Change in resting heart rate
Change from baseline blood pressure | with 2 month
  Change in systolic blood pressure

IPD SHARING:
Plan to Share IPD: Undecided